CLINICAL TRIAL: NCT00127387
Title: A Prospective, Randomized Pilot Study of Enbrel VS Placebo in Patients Receiving Radiation Therapy to Combat Fatigue and Cachexia
Brief Title: Enbrel Versus Placebo With Radiation Therapy to Combat Fatigue and Cachexia
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: PI moved to Oregon
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Sanchez Cancer Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 001-0015-211
Record Dates: First submitted 2005-08-03; First posted 2005-08-05 (Estimated); Last update posted 2012-06-26 (Estimated); Status verified 2012-06

CONDITIONS: Lung Cancer; Prostate Cancer; Neoplasm Metastasis; Bone Cancer
Keywords: Bone metastasis; Radiation therapy; Lung cancer; Prostate cancer; Advanced lung cancer receiving radiation therapy; Advanced prostate cancer receiving radiation therapy; Any cancer with bone mets receiving radiation therapy
MeSH Terms: conditions — Lung Neoplasms; Prostatic Neoplasms; Neoplasm Metastasis; Bone Neoplasms | interventions — Etanercept

INTERVENTIONS:
Drug: Enbrel

SUMMARY:
Patients who receive radiation therapy often have fatigue or a decrease in feeling well causing a "wasting" away. For patients with advanced disease of lung cancer, prostate cancer, or cancer that has spread to the bone, it is hoped that this drug may decrease this. If patients feel better during treatments they can complete the therapy without any breaks in treatment. For treatment to be most effective, it should be given in the amount needed, on a particular schedule.

DETAILED DESCRIPTION:
Subjects will be placed in a group to receive either the drug enbrel, or a placebo. The radiation therapy treatments are as they would be given if the person was not on a research study. The selection of the group a patient is in is done by random, like flipping a coin. The doctor is not able to influence which group anyone is selected for. As is done routinely, radiation therapy is given Monday through Friday for about 4 to 6 weeks.The injections of enbrel or placebo are given two times a week. The enbrel or placebo is given as an injection directly under the skin with a small needle.

ELIGIBILITY:
Inclusion Criteria:

* Advanced lung, prostate, or bony metastasis for cancer
* Performance status (PS) of 3 or less
* Good lab test results with albumin of at least 2.5
* Radiation therapy of at least 4000Gy in 4 weeks

Exclusion Criteria:

* Poor PS
* Planned radiation therapy for less than 4 weeks or 4000Gy
* Limited disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2001-05; Primary Completion 2005-09 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Determine if the subjects who received the enbrel study drug had a better quality of life than the subjects who received placebo

SECONDARY OUTCOMES:
Safety profile for enbrel taken by this group of individuals

CONTACTS AND LOCATIONS:
Overall Officials: Charles R Thomas, Jr, MD, Principal Investigator — U Texas Health Science Center San Antonio
Locations (1):
- University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States